CLINICAL TRIAL: NCT01954212
Title: A Multi-centred, Stepped Wedge, Cluster Randomised Controlled Trial to Compare the Clinical and Cost Effectiveness of a Complex Oral Health Care Intervention and Standard Oral Health Care in Stroke Care Settings: a Phase II Pilot Trial.
Brief Title: Stroke Oral healthCare pLan Evaluation
Acronym: SOCLE II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: Nursing Midwifery and Allied Health Profession (NMAHP) Research Unit (Unknown); University of Glasgow (Other); NHS Lanarkshire (Other Government); Glasgow Dental Hospital and School (Unknown); University of Edinburgh (Other)
Responsible Party: Principal Investigator, Prof. Marian Brady, Professor, Glasgow Caledonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TSA 2012/09
Record Dates: First submitted 2013-08-21; First posted 2013-10-01 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Cerebrovascular Disorders; Stroke; Pneumonia; Oral Hygiene
Keywords: Oral health
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke; Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced complex oral health care intervention (Experimental): The complex oral health care (OHC) intervention (SOCLE intervention) includes patient, staff and service level interventions.
  Interventions: Other: Enhanced complex oral health care
- Usual oral health care (No Intervention): Oral health care (OHC) will be provided in the standard manner, with no change to usual care.
  Provision of this standard OHC will be sampled monthly. Surveys suggest that standard oral health care (OHC) in stroke care settings comprise poorly supported OHC interventions delivered by staff that lacked access to specialist training, products, equipment, assessments, protocols and dental services.

INTERVENTIONS:
Other: Enhanced complex oral health care — Our proposed complex oral health care (OHC) intervention (SOCLE intervention) comprises 3 levels of intervention:
  1. Patient Level: An individualised OHC assessment on admission and individualised OHC plans for patients, which may involve staff-led OHC support, access to OHC equipment, products and specialist support services and OHC health promotion components.
  2. Staff Level: Specialist web-based OHC educational training, including information on the oral cavity and structures; oral health problems (e.g. decay, gum disease, dry mouth); instruction on OHC techniques, equipment and products; use of the SOCLE assessment and protocol tools.
  3. Service Level: Processes to facilitate access to specialist dental support services (e.g. dentist, hygienist, denture repair laboratory). Essential OHC equipment (toothbrushes, denture marking kits) and products (e.g. toothpaste, oral balance gel) on the ward will be available.
  Arms: Enhanced complex oral health care intervention

SUMMARY:
Stroke associated pneumonia (SAP) affects a fifth of stroke survivors annually, tripling the risk of death at 30 days and contributing to poorer rehabilitation outcomes, prolonged hospital stays and dependency at discharge. Systematic review evidence indicates that enhanced oral health care (OHC) has a preventative effect on the incidence of pneumonia amongst nursing home populations (absolute risk reductions 6.6% to 11.7%; numbers needed to treat 8.6 to 15.3 individuals). There are strong theoretical reasons to suggest similar benefits might be observed in stroke care settings but current empirical evidence is weak - trial quality (randomisation, blinding, sample size, reporting), intervention description and thus feasibility of translation into clinical practice is very poor. Following an extensive pre-clinical programme of work, investigators now plan the pilot phase (Phase II) of a stepped-wedge cluster RCT of a well-developed and defined complex OHC intervention versus usual OHC. Investigators aim to establish a robust web-based randomisation process, refine the proposed intervention (training, tools, equipment), recruitment, adherence, record linkage and sampling methodologies. Investigators also aim to establish the relationship between SAP and plaque and any diversity between sites.

DETAILED DESCRIPTION:
SOCLE II is the pilot phase (Phase II) of a stepped-wedge cluster randomised controlled trial (RCT) of a complex oral health care (OHC) intervention versus usual OHC.

SOCLE II aims to evaluate the feasibility of a full scale pragmatic trial of the clinical and cost effectiveness of a complex OHC package of care versus usual care for people in stroke care settings. Ward level cluster randomisation will progress in a stepped wedge manner where after a period of baseline data collection each ward in a randomly allocated order will 'convert' from usual care to an enhanced oral health care intervention.

This pilot trial will assess the feasibility of delivering this enhanced OHC intervention across four sites and will inform the trial design of a full scale phase III trial including refining the proposed intervention (training, tools, equipment), recruitment, adherence, record linkage, sampling methodologies, sample size calculations and pilot our health economic evaluation. Investigators also aim to establish the relationship between SAP and plaque and any diversity between sites. Our proposed pilot work will support an application for a planned Phase III definitive trial.

Principal Research Questions:

(i) Are the SOCLE intervention and data collection process viable across multiple sites? (ii) Can sample size calculations and estimates of recruitment and retention be refined? (iii) Can pneumonia event rates across several sites and distribution over time post stroke onset be determined? (iv) Can the association between dental and denture plaque and SAP be established? (v) Can the predetermined criteria for progression to Phase III definitive multi-centred stepped wedge cluster RCT with economic evaluation be met?

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to stroke care settings.

Exclusion Criteria:

* Consent declined.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pneumonia | Weekly assessments for the duration of ward stay until discharge, an expected average stay of no more than 3 weeks.
  Based on the Mann Criteria for Chest infection and evaluated based on concurrent review of case notes at each weekly data collection point and a retrospective review of case notes on discharge.

SECONDARY OUTCOMES:
Oral Health Impact Profile | Weekly assessments for the duration of ward stay until discharge, an expected average stay of no more than 3 weeks.
  Patient rated Oral Health Impact Profile (with activity and participation components, Locker et al 2002)
Dental plaque | Weekly assessments for the duration of ward stay until discharge, an expected average stay of no more than 3 weeks.
Denture plaque | Weekly assessments for the duration of ward stay until discharge, an expected average stay of no more than 3 weeks.
Antibiotics prescribed | Weekly for the duration of ward stay until discharge, an expected average stay of no more than 3 weeks.
  The prescription of antibiotics and type of antibiotic prescription will be documented from the drug kardex.
Death | Participants will be followed for the duration of hospital stay, an expected average stay of no more than 3 weeks.

OTHER OUTCOMES:
Length of hospital stay | Determined at point of discharge from hospital ward (expected average stay of no more than 3 weeks).
Discharge destination | Determined at point of discharge from hospital ward (expected average stay of no more than 3 weeks).
Knowledge and attitudes of staff | 1. Prior to OHC training package (3 to 10 months after start of recruitment depending on randomised allocation). 2. After completion of training package. 3. At close of study (16 months after recruitment starts at the initial site).
  In this stepped-wedge randomised controlled trial design staff will be asked to complete knowledge and attitudes questionnaires (Frenkel 2001) at the 3 stated time points. (Ref: Frenkel HF et al. Improving oral health of institutionalised elderly people by educating caregivers. Community Dent Oral Epidemiol 2001;29:289-97)
Adherence | Weekly assessments for the duration of study (16 months).
  Adherence to study protocol - including completed assessments, documented oral health care plans
OHC resource use | Weekly assessments for the duration of study (16 months).
  Oral health care equipment and product resource use questionnaire, and specialist services resource use questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marian Brady, Principal Investigator — Glasgow Caledonian University
Locations (4):
- United Kingdom (4):
  - Hairmyres Hospital, East Kilbride, Lanarkshire
  - Wishaw General Hospital, Wishaw, Lanarkshire
  - Stobhill Hospital, Glasgow, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland

REFERENCES:
- [Derived] Brady MC, Stott DJ, Weir CJ, Chalmers C, Sweeney P, Barr J, Pollock A, Bowers N, Gray H, Bain BJ, Collins M, Keerie C, Langhorne P. A pragmatic, multi-centered, stepped wedge, cluster randomized controlled trial pilot of the clinical and cost effectiveness of a complex Stroke Oral healthCare intervention pLan Evaluation II (SOCLE II) compared with usual oral healthcare in stroke wards. Int J Stroke. 2020 Apr;15(3):318-323. doi: 10.1177/1747493019871824. Epub 2019 Sep 30. PMID 31564241
- [Derived] Brady MC, Stott D, Weir CJ, Chalmers C, Sweeney P, Donaldson C, Barr J, Barr M, Pollock A, McGowan S, Bowers N, Langhorne P. Clinical and cost effectiveness of enhanced oral healthcare in stroke care settings (SOCLE II): a pilot, stepped wedge, cluster randomized, controlled trial protocol. Int J Stroke. 2015 Aug;10(6):979-84. doi: 10.1111/ijs.12530. Epub 2015 Jun 16. PMID 26079661